CLINICAL TRIAL: NCT04944121
Title: A Phase 2, Double-blind, Placebo-controlled Study of RSLV-132 in Subjects With Post-acute COVID-19 (Long COVID)
Brief Title: Phase 2 Study of RSLV-132 in Subjects With Long COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resolve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132-05
Record Dates: First submitted 2021-06-25; First posted 2021-06-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2022-11

CONDITIONS: Post-acute Corona Virus 19 (COVID-19) (Long COVID)
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — RSLV-132; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSLV-132 (Experimental): RSLV-132 is an enzymatically active ribonuclease designed to digest the ribonucleic acid contained in autoantibodies and immune complexes and thereby render them biologically inert. A dose of 10 mg/kg will be administered by intravenous infusion on Days: 1, 8, 15, 29, 43, and 57
  Interventions: Drug: RSLV-132
- Placebo (Placebo Comparator): Sodium chloride 0.9% will be administered by intravenous infusion on Days: 1, 8, 15, 29, 43, and 57
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: RSLV-132 — 10 mg/kg RSLV-132 administered by intravenous infusion
  Arms: RSLV-132
Drug: Sodium Chloride 0.9% — 0.9% sodium chloride administered by intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy (decrease in profound fatigue), safety and pharmacokinetics of RSLV-132 in subjects with long Corona Virus (COVID) syndome

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled study in approximately 70 subjects with long COVID syndrome. After being informed about the study and potential risks, all subjects giving written informed consent will be screened to determine eligibility in the 21 days before the start of study treatment. Prior to the first study treatment administration, subjects will be randomized in a 2:1 ratio to receive six administrations of 10 mg/kg RSLV-132 or placebo on Days 1, 8, 15, 29, 43 and 57. Subjects will then attend an end of study visit approximately 10 weeks after the start of treatment (Day 71).

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by qualitative Polymerase Chain Reaction (PCR) at least 24 weeks prior to Baseline
* PROMIS Fatigue SF 7a raw score of 21 or greater at Screening (confirm onset of fatigue was post-infection)
* Able to communicate and able to provide valid, written informed consent
* Ages 18 to 75 inclusive
* Minimum weight of 45 kg
* Female participants shall be either of non-child-bearing potential (permanently sterilized by bilateral tubal occlusion, hysterectomy, or bilateral salpingectomy), or menopausal (more than one year since last menstrual cycle and confirmed by blood FSH levels > 22 mIU/mL) OR practicing highly effective contraception (e.g., oral (but not including progestogen-only oral contraceptives), injectable, implantable or transdermal contraceptives, a non-hormonal intrauterine device [IUD] or an intrauterine hormone releasing system [IUS]) for at least 2 months prior to dosing and until 125 days after the last dose. In terms of sexual relations, female participants not practicing highly effective contraception as described above should abstain or only engage with male partners who are sterile or vasectomized. Female participants of child-bearing potential will also be required to have a negative serum pregnancy test [beta human chorionic gonadotropin [ß-hCG]) at Screening and negative pregnancy urine test at Baseline. Female participants must agree not to donate eggs from the first dose until 125 days after the last dose
* Male participants, who are not sterile or vasectomized, must agree to abstain or only engage with female partners who use highly effective contraception from the first dose until 125 days after the last dose. Male participants must also agree not to donate sperm from the first dose until 125 days after the last dose

Exclusion Criteria:

* Previous admission to the intensive care unit for COVID-19-related symptoms
* Presence of orthostatic hypotension or tachycardia at Screening
* Completion of COVID-19 vaccination less than 4 weeks of Baseline (i.e., 4 weeks after the second dose of a two-dose vaccine or 4 weeks after a single dose vaccine)
* Use of therapies to treat COVID-19 symptoms such as remdesivir, dexamethasone (or any other corticosteroid), or convalescent plasma within 14 days of Baseline
* Use of concomitant medications that are sedating
* Screening lab abnormalities that may cause fatigue such as severe anemia or hypocalcaemia
* History of anaphylaxis to a medication, diet, or environmental exposure such as bee sting
* Previous diagnosis of chronic fatigue syndrome, fibromyalgia, lupus, Sjogren's syndrome, or postural orthostatic tachycardia syndrome (POTS)
* Previous diagnosis of sleep apnea
* Participation in another clinical study with receipt of an investigational product within 3 months or 5 half- lives, of last administration (whichever is longer) from Baseline
* The presence of a clinically significant infection in the judgement of the Investigator, within seven days of Baseline
* Positive test for hepatitis B, C, or HIV at Screening
* Positive pregnancy test at Screening or Baseline
* Female subjects currently pregnant or breast feeding at Baseline
* Inability or unwillingness to comply with protocol-specified procedures which, in the opinion of the Investigator, would make the subject unsuitable for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
PROMIS Fatigue SF 7a T-score | From Baseline to Day 71
  Mean change in Patient-Reported Outcomes Measurement Information System Fatigue Short Form 7a (PROMIS Fatigue 7a) T-score at the end of treatment compared to baseline. The PROMIS Fatigue 7a consists of seven questions measuring symptoms severity at five-point intervals, with higher scores representing a worse outcome.

SECONDARY OUTCOMES:
FACIT Fatigue questionnaire | From Baseline to Day 71
  Comparison of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire at the end of treatment compared to baseline. The FACIT-F is a 13 item measure of fatigue with a 7 day recall memory. Items are scored on a five point scale (0-not at all to 4-very much). The total score therefore ranges from 0 to 52, with higher scores reflecting greater fatigue.
Long COVID-19-related Symptom Assessment patient questionnaire | From Baseline to Day 71
  Comparison of the Long COVID-19-related Symptom Assessment patient questionnaire at the end of treatment compared to baseline. Subjects will be asked to describe the severity of eight COVID-19 related symptoms (muscle pain, joint pain, chest pain, brain fog, chills, sweats, abdominal pain and chest tightness) over the last 7 days on a four point scale (0-none to 3-severe) with a higher score representing a worse outcome.
Patient-reported Global Impression of Severity questionnaire | From Baseline to Day 71
  Comparison of the Patient-reported Global Impression of Severity (PGIS) questionnaire at the end of treatment compared to baseline. Subjects will be asked to describe the severity of fatigue on the assessment day compared to the past 7 days on a four point scale (1-no improvement to 4-significant improvement) with a higher score representing a better outcome.
Digit Symbol Substitution Test | From Baseline to Day 71
  Comparison of the Digit Symbol Substitution Test (DSST) at the end of treatment compared to baseline. The DSST is a highly validated measure of the patient's ability to focus and concentrate of a simple task. Subjects with profound fatigue take more time to complete the test.
Physician Global Assessment | From Baseline to Day 71
  Comparison of the Physician Global Assessment at the end of treatment compared to baseline. The assessment is measured on a 0 to 100 mm scale with score 0 to be no disease activity and score 100 to be the most severe disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: James Posada, Study Director — Resolve Therapeutics LLC
Locations (5):
- United States (5):
  - Resolve Clinical Center, Mobile, Alabama
  - Resolve Clinical Center, Coral Gables, Florida
  - Resolve Clinical Center, Pompano Beach, Florida
  - Resolve Clinical Center, Knoxville, Tennessee
  - Resolve Clinical Center, Seattle, Washington